CLINICAL TRIAL: NCT02250781
Title: A First-in-Human Phase I Single-Agent Open-Label Dose-Escalation Study of Every Three-Week Dosing of Oral ONC201 in Patients With Advanced Solid Tumors
Brief Title: Oral ONC201 in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Rutgers Cancer Institute of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 051403; NCI-2014-01305 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 051403 (Other: Rutgers Cancer Institute of New Jersey); P30CA072720 (NIH)
Record Dates: First submitted 2014-07-28; First posted 2014-09-26 (Estimated); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Solid Tumors
MeSH Terms: interventions — TIC10 compound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Oral ONC201) (Experimental): Patients receive Oral ONC201 PO on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Oral ONC201

INTERVENTIONS:
Drug: Oral ONC201 — Given PO
  Other Names: ONC201; TIC10

SUMMARY:
This phase I trial studies the side effects and best dose of Oral ONC201 in treating patients with advanced solid tumors. Oral ONC201 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the recommended phase II dose of single agent ONC201 orally once every three weeks.

SECONDARY OBJECTIVES:

I. To characterize pharmacokinetics of ONC201. II. To assess serum biomarkers of therapeutic response to ONC201. III. To assess preliminary antitumor activity of ONC201 as a single agent in advanced solid tumors.

OUTLINE: This is a dose-escalation study.

Patients receive ONC201 orally (PO) on day 1. Courses repeat every 21 days for a total of 2 courses.

After completion of study treatment, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an advanced solid tumor that is refractory to standard treatment, or for which no standard therapy is available, or the subject refuses standard therapy
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1
* All patients must have measurable or evaluable disease defined by Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 criteria; if the patient has received prior radiation therapy one measurable lesion must be outside the irradiated field; lesions within an irradiated field will be followed as non-target lesions and considered evaluable; if the only site of measurable disease is within a previously irradiated field then 6 months must have elapsed between the completion of radiation therapy and entry on study to be considered measurable
* Patients are eligible for enrollment if they have not had prior investigational or approved cytotoxic chemotherapy within 28 days prior to the first dose (week 1, day 1); 42 days in the case of alkylating agents; 28 days or 5 half-lives (whichever is less; but not less than 14 days) in case of investigational or approved molecularly targeted agent; 14 days in the case of radiotherapy; any number of prior therapies is allowable
* All adverse events grade =< 2 related to prior therapies (chemotherapy, radiotherapy, and/or surgery) must be resolved, except for alopecia or neuropathy; patients are eligible for enrollment if they have had no surgery in the prior 6 weeks (minor surgical procedures such as skin biopsies and port placement done on an outpatient basis do not require a waiting period)
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9.0 mg/dL without transfusion in 2 prior weeks
* Total bilirubin within normal range; for patients with liver metastases, serum bilirubin =< 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate transaminase [SGPT]) =< 2.5 x upper limit of normal
* Measured OR estimated creatinine clearance >= 40 mL/min/1.73 m^2 for patients with creatinine levels above normal
* Men or women treated or enrolled on this protocol must agree to use double barrier contraceptives; oral, implantable, or injectable contraceptives are not considered effective for this study; women of child-bearing potential must have a negative serum pregnancy test =< 72 hours prior to initiating treatment; subjects must agree to use double barrier contraceptive therapy for the duration of study participation, and 4 months after completion of ONC201 administration; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Tumor specimen (paraffin-embedded block or frozen tissue) from prior resection or biopsy available that is sufficient to perform pharmacodynamic assays (>= 3 slides for immunohistochemistry [IHC]) - mandatory for patients in the dose expansion cohort only
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients with symptomatic brain metastases are excluded; however, patients with asymptomatic central nervous system (CNS) metastases may participate in this trial; the patient must have completed any prior local treatment for CNS metastases > 28 days prior to study entry including radiotherapy or surgery; patients receiving steroids for CNS metastases may not participate on this study
* Prior bevacizumab for treatment of glioblastoma or high grade glioma
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ONC201 or its excipients
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements
* Patient is unable or unwilling to abide by the study protocol or cooperate fully with the investigator
* Patients with a known human immunodeficiency virus (HIV)-positive test on combination antiretroviral therapy are ineligible for the initial first-in-man trial
* Patient has active cardiac disease including any of the following:

  * Corrected QT (QTc) > 500 msec on screening electrocardiogram (ECG) (using the QTc Fridericia [F] formula)
  * Angina pectoris that requires the use of anti-anginal medication
  * Ventricular arrhythmias except for benign premature ventricular contractions
  * Supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medication
  * Conduction abnormality requiring a pacemaker
  * Valvular disease with document compromise in cardiac function
  * Symptomatic pericarditis
* Patient has a history of cardiac dysfunction including any of the following:

  * Myocardial infraction within the last 6 months, documented by persistent elevated cardiac enzymes or persistent regional wall abnormalities on assessment of left ventricular ejection fraction (LVEF) function
  * History of documented congestive heart failure (New York Heart Association functional classification III-IV)
  * Documented cardiomyopathy
* Patient with stroke in the last 3 months
* Patients with a history of seizures with in the past 3 months
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of ONC201 (uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
* Patients who have been treated with any hematopoietic colony-stimulating growth factors (e.g., filgrastim [G-CSF], granulocyte-macrophage colony-stimulating factor [GM-CSF]) =< 2 weeks prior to starting study drug; erythropoietin or darbepoetin therapy, if initiated at least 2 weeks prior to enrollment, may be continued
* Women who are pregnant or breast feeding or adults of reproductive potential not employing an effective method of birth control; double barrier contraceptives must be used through the trial by both sexes; oral, implantable, or injectable contraceptives are not considered effective for this study
* Women of child-bearing potential must have a negative serum pregnancy test =< 72 hours prior to initiating treatment
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, must use highly effective contraception during treatment and for 16 additional weeks after stopping treatment; the highly effective contraception is defined as either:

  * True abstinence: when this is in line with the preferred and usual lifestyle of the subject; periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
  * Sterilization: have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago; in case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
  * Male partner sterilization (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate); for female subjects on the study, the vasectomized male partner should be the sole partner for that patient
  * Use of a combination of any two of the following (a+b):

    1. Placement of an intrauterine device (IUD) or intrauterine system (IUS)
    2. Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository
  * Oral contraception, injected or implanted hormonal methods are not allowed
  * Fertile males, defined as all males physiologically capable of conceiving offspring must use condom during treatment and for an additional 16 weeks after stopping treatment
  * Female partner of male study subject should use highly effective contraception during dosing of any study agent and for 16 weeks after final dose of study therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2015-01-12 (Actual); Primary Completion 2018-10-18 (Actual); Study Completion 2018-10-25 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity rate during cycle 1 of treatment with oral ONC201 | Day 21

SECONDARY OUTCOMES:
Recommended phase II dose (RP2D) for oral ONC201 | At the end of 6 weeks therapy
Frequency of toxicities associated with ONC201 | Up to 4 weeks after end of study treatment
Pharmacokinetics of oral ONC201 - Half-life | Up to 4 weeks of therapy
Pharmacokinetics of oral ONC201 - Maximum concentration | Up to 4 weeks of therapy
Pharmacokinetics of oral ONC201 - Area under the curve (AUC) over time | Up to 4 weeks of therapy
Response rate of oral ONC201 in patients with advanced solid tumors | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jyoti Malhotra, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey, United States

REFERENCES:
- [Derived] Stein MN, Malhotra J, Tarapore RS, Malhotra U, Silk AW, Chan N, Rodriguez L, Aisner J, Aiken RD, Mayer T, Haffty BG, Newman JH, Aspromonte SM, Bommareddy PK, Estupinian R, Chesson CB, Sadimin ET, Li S, Medina DJ, Saunders T, Frankel M, Kareddula A, Damare S, Wesolowsky E, Gabel C, El-Deiry WS, Prabhu VV, Allen JE, Stogniew M, Oster W, Bertino JR, Libutti SK, Mehnert JM, Zloza A. Safety and enhanced immunostimulatory activity of the DRD2 antagonist ONC201 in advanced solid tumor patients with weekly oral administration. J Immunother Cancer. 2019 May 22;7(1):136. doi: 10.1186/s40425-019-0599-8. PMID 31118108